CLINICAL TRIAL: NCT05811455
Title: Comparative Effects of Aerobic Exercises and Progressive Muscle Relaxation Exercises on Pain,Anxiety and Quality of Life
Brief Title: Comparative Effects of Aerobic Exercises and Progressive Muscle Relaxation Exercises on Pain and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/054
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Pain Syndrome; Anxiety
MeSH Terms: conditions — Somatoform Disorders; Anxiety Disorders | interventions — Exercise; Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: aerobic exercises. (Experimental): The first treatment group will be given aerobic exercises for six weeks at least three times per week. This group will include 14 participants. This study group will be assigned with basic treatment protocol with aerobic exercises along with 10 minutes of warm up period.
  Interventions: Other: Aerobic exercises
- group b progressive muscle relaxation exercises. (Active Comparator): The intervention will be given three days per week for six weeks. Pre and post-treatment readings will be noted. Each total session will last for 45 minutes. The importance of the study will be explained, and consent will be taken from the people before the intervention will be applied.
  * Breathe in, and tense the first muscle group (hard but not to the point of pain or cramping) for 4 to 10 seconds.
  * Breathe out, and suddenly and completely relax the muscle group (do not relax it gradually) (20)
  Interventions: Other: Progressive muscle relaxation
- Group C. Control group (No Intervention): No intervention was given

INTERVENTIONS:
Other: Aerobic exercises — To compare the effects of aerobic exercise and progressive muscle relaxation exercises on pain and quality of life in premenstrual syndrome
  Arms: Group A: aerobic exercises.
Other: Progressive muscle relaxation — progressive muscle relaxation exercises.
  Arms: group b progressive muscle relaxation exercises.

SUMMARY:
Premenstrual syndrome is the clinical condition in which reproductive age females suffer from emotional and physical symptoms not related to any disease, starting usually 5 days before the menstrual cycle for 3 consecutive cycles.

DETAILED DESCRIPTION:
Premenstrual syndrome is the clinical condition in which reproductive age females suffer from emotional and physical symptoms not related to any disease, starting usually five days before the menstrual cycle for three consecutive cycles. As menstrual cycle starts in females these symptoms vanish on 4th day of menstruation. Around 10% to 53% of female adults suffer from this condition. This condition limits activities of daily life and adversely effects the quality of life therefore, the administration of proper medical intervention is very important. Aerobic exercises and progressive muscle relaxation exercises have been effective in the treatment of premenstrual syndrome previously in a few studies. However, these two interventions have never been compared to test their effects on pain, and functional performance.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 40 years
* Females in their last week of the luteal phase (1 week before menstruation)
* Females with regular menstrual with equal intervals between 21 and 35 days
* Females with a score of 133 and above after being screened with Premenstrual syndrome scale
* Females suffering from PMS for at least the past six months

Exclusion Criteria:

* Females with the irregular menstrual cycle
* Pregnant females
* Menstruating females or females in the follicular or ovulatory phase
* History of physical exercise in the past three months before the beginning of the study
* Females suffering from other gynecological issues such as endometriosis, PCOS, uterine or cervical cancer

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
1. For Anxiety, Depression: • DASS-21 The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) | 6 weeks
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress.(16)
Numerical rating scales (NRSs) | 6 weeks
  Numerical rating scales (NRSs) are the simplest and most commonly used scale. The numerical scale is most commonly 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable
• SF-36 The 36-Item Short Form Health Survey questionnaire (SF-36) | 6 weeks
  The 36-Item Short Form Health Survey questionnaire (SF-36) is a very popular instrument for evaluating Health-Related Quality of Life. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH)

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Tariq, Mphill, Principal Investigator — Riphah International University
Locations (1):
- Johar Institute of Professional Studies, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No